CLINICAL TRIAL: NCT00827528
Title: Surgical Treatment of Anterior Vaginal Wall Prolapse: Comparison of SIS Graft and Traditional Repair.
Brief Title: SIS Graft and Traditional Repair in Vaginal Wall Prolapse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Paulo Cezar Feldner Jr, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SISAPI 01
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; Surgical Treatment
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SIS graft (Experimental): this group will use a biologic graft (SIS - Small Intestine Submucosa) in correction of anterior vaginal wall prolapse.
  Interventions: Procedure: Biologic Graft (SIS)
- 2 (Active Comparator): this group will use a traditional repair on correction of anterior vaginal wall prolapse.
  Interventions: Procedure: Traditional correction of anterior vaginal wall prolapse

INTERVENTIONS:
Procedure: Traditional correction of anterior vaginal wall prolapse — Traditional repair.
  Patients diagnosed with anterior vaginal wall prolapse will be submitted to surgical correction. They will be randomized to receive a traditional repair or a graft in surgery.
  Arms: 2
Procedure: Biologic Graft (SIS) — Biologic graft (SIS - Small Intestine Submucosa) in correction of anterior vaginal wall prolapse.
  Patients diagnosed with anterior vaginal wall prolapse will be submitted to surgical correction. They will be randomized to receive a traditional repair or a graft in surgery.
  Arms: SIS graft

SUMMARY:
The objective of this study is to evaluate surgical treatment of anterior vaginal wall prolapse using the sis graft or traditional repair. This a randomized and prospective study. Clinical patterns that will be evaluated: anatomic results of surgery; impact of surgery in quality of life using the Pelvic Organ Prolapse Questionnaire (P-QoL), sexual function with FSFI and possible complications.

DETAILED DESCRIPTION:
The objective of this study is to evaluate surgical treatment of anterior vaginal wall prolapse using the sis graft or traditional repair. This a randomized and prospective study. Clinical patterns that will be evaluated: anatomic results of surgery; impact of surgery in quality of life using the Pelvic Organ Prolapse Questionnaire (P-QoL), sexual function with FSFI and possible complications

ELIGIBILITY:
Inclusion Criteria:

* anterior vaginal wall prolapse with poin Ba at least at +1;
* pre and postmenopausal patients

Exclusion Criteria:

* patients without surgical indication;
* infection;
* coagulopathy;
* gynecologic cancer;
* liver or kidney active diseases.

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
surgical anatomic results | one year

SECONDARY OUTCOMES:
impact on quality of life using the Pelvic Organ Prolapse Questionnaire (P-QoL); sexual function with FSFI; complications | one year

CONTACTS AND LOCATIONS:
Overall Officials: Manoel João BC Girão, PhD, Study Chair — Department of Gynecology, Federal University of São Paulo; Paulo C Feldner Jr, MD, Principal Investigator — Department of Gynecology, Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo/SP, Brazil

REFERENCES:
- [Result] Sung VW, Rogers RG, Schaffer JI, Balk EM, Uhlig K, Lau J, Abed H, Wheeler TL 2nd, Morrill MY, Clemons JL, Rahn DD, Lukban JC, Lowenstein L, Kenton K, Young SB; Society of Gynecologic Surgeons Systematic Review Group. Graft use in transvaginal pelvic organ prolapse repair: a systematic review. Obstet Gynecol. 2008 Nov;112(5):1131-42. doi: 10.1097/AOG.0b013e3181898ba9. PMID 18978116
- [Result] Bako A, Dhar R. Review of synthetic mesh-related complications in pelvic floor reconstructive surgery. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jan;20(1):103-11. doi: 10.1007/s00192-008-0717-5. Epub 2008 Sep 9. PMID 18779916
- [Result] Jia X, Glazener C, Mowatt G, MacLennan G, Bain C, Fraser C, Burr J. Efficacy and safety of using mesh or grafts in surgery for anterior and/or posterior vaginal wall prolapse: systematic review and meta-analysis. BJOG. 2008 Oct;115(11):1350-61. doi: 10.1111/j.1471-0528.2008.01845.x. Epub 2008 Aug 19. PMID 18715243
- [Result] Maher C, Baessler K, Glazener CM, Adams EJ, Hagen S. Surgical management of pelvic organ prolapse in women: a short version Cochrane review. Neurourol Urodyn. 2008;27(1):3-12. doi: 10.1002/nau.20542. PMID 18092333
- [Result] Chen CC, Ridgeway B, Paraiso MF. Biologic grafts and synthetic meshes in pelvic reconstructive surgery. Clin Obstet Gynecol. 2007 Jun;50(2):383-411. doi: 10.1097/GRF.0b013e31804b184c. PMID 17513926
- [Result] Silva WA, Karram MM. Scientific basis for use of grafts during vaginal reconstructive procedures. Curr Opin Obstet Gynecol. 2005 Oct;17(5):519-29. doi: 10.1097/01.gco.0000180156.64879.00. PMID 16141767
- [Result] Maher C, Baessler K, Glazener CM, Adams EJ, Hagen S. Surgical management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD004014. doi: 10.1002/14651858.CD004014.pub3. PMID 17636742
- [Result] Maher C, Baessler K. Surgical management of anterior vaginal wall prolapse: an evidencebased literature review. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Feb;17(2):195-201. doi: 10.1007/s00192-005-1296-3. Epub 2005 May 25. PMID 15915320